CLINICAL TRIAL: NCT02482441
Title: A Phase 1a/b Dose Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of OMP-131R10 in Advanced Solid Tumors and in Combination With FOLFIRI for Patients With Previously Treated Metastatic Colorectal Cancer
Brief Title: A Phase 1a/b Dose Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of OMP-131R10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 131R10-001
Record Dates: First submitted 2015-06-19; First posted 2015-06-26 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Advanced Relapsed Tumors; Refractory Solid Tumors
Keywords: Advanced Solid Tumors and in Combination; FOLFIRI for Patients with Previously Treated Metastatic; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMP-131R10 intravenous (in the vein) infusions (Experimental): OMP-131R10 will be administered IV on the first day of each 14-day cycle.
  Interventions: Drug: OMP-131R10; Drug: FOLFIRI
- FOLFIRI (5-FU, irinotecan, leucovorin). (Experimental): dosing continues up to the 20 mg/kg dose level
  Interventions: Drug: OMP-131R10; Drug: FOLFIRI

INTERVENTIONS:
Drug: OMP-131R10 — There are 5 planned dose cohorts of OMP-131R10. Dose escalation will follow a traditional 3+3 framework. Treatment will be continued until progressive disease or unacceptable toxicity.
  Other Names: OMP-131R10, IgG1 humanized monoclonal antibody
Drug: FOLFIRI — Treatment will consist of OMP-131R10 and the FOLFIRI chemotherapy regimen.

SUMMARY:
This is an open-label Phase 1a/b dose-escalation study to assess the safety, tolerability, and PK of OMP-131R10 as a single agent for advanced solid tumors and in subjects with metastatic colorectal cancer.

DETAILED DESCRIPTION:
The Phase 1a portion of the study in subjects with advanced solid tumors will consist of a dose escalation part followed by a dose-expansion cohort. OMP-131R10 will be administered IV on the first day of each 14-day cycle.

Dose escalation will follow a traditional 3+3 framework. Treatment will be continued until progressive disease or unacceptable toxicity.

The Phase 1b portion of the study will be conducted in subjects with metastatic colorectal cancer whose tumors have progressed after at least 1 line of therapy for metastatic disease.

Treatment will consist of OMP-131R10 and the FOLFIRI chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for the study:

1. Phase 1a portion: Histologically confirmed advanced relapsed or refractory solid tumors that have exhausted standard of care therapy or either refuse or are not considered to be candidates for any remaining standard therapy.
2. Age ≥18 years
3. ECOG performance status 0 or 1 (see Appendix B)
4. Must have evaluable disease per RECIST 1.1. (see Appendix C)
5. Subjects must have Formalin-Fixed, Paraffin-Embedded (FFPE) tissue available either archived or fresh core or punch needle biopsied at study entry (two fresh cores/punches preferred whenever possible).
6. Must have received their last anti-cancer therapy, including radiotherapy, chemotherapy, biologic therapy, or herbal therapy at least 3 weeks or 5 half-lives (for systemic agents), whichever is shorter, from initiation of study treatment.
7. Platelets >100,000/mL without transfusions in the past 7 days
8. Total bilirubin within 1.5x institutional upper limit of normal (ULN)

   * AST (SGOT) and ALT (SGPT) <3 X institutional ULN
   * Patients with documented liver metastases: AST (SGOT) and/or ALT (SGPT) ≤ 5 × ULN
   * Albumin ≥ 3.0 g/dL
   * Creatinine <1.5 X institutional ULN OR
   * Creatinine clearance >50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Currently receiving any therapeutic treatment for their malignancy including other investigational agents
2. Uncontrolled seizure disorder, active neurologic disease, or active CNS involvement except for individuals who have previously treated CNS metastases, are asymptomatic, and have no requirement for a corticosteroid dose (indicated to reduce brain edema) that is equivalent to a prednisone dose of >10mg orally per day or anti-seizure medication for at least 4 weeks prior to first dose of study drug.
3. History of a Grade 3 or 4 allergic reaction attributed to humanized or human monoclonal antibody therapy
4. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant women or nursing women
6. Subjects with congestive heart failure with New York Heart Association Classification III, or IV (see Appendix D)
7. Known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07-16 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | DLTs during the evaluation (28 days)
  Subject will be assessed for DLTs during the evaluation window (28 days). Once the maximum tolerated dose (MTD) or maximum administered dose (MAD) has been determined.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - UCSF, San Francisco, California
  - University of Colorado Hospital Anschulz Cancer Pavilion, Aurora, Colorado
  - Yale, New Haven, Connecticut
  - Massachusetts General Hospital, Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - M.D. Anderson Cancer Center, Houston, Texas